CLINICAL TRIAL: NCT02941991
Title: Follow-up to 5 Years of a Phase I/II, Open-Label, Multi-Center, Prospective Study to Determine the Safety and Tolerability of Sub-retinal Transplantation of Human Embryonic Stem Cell Derived Retinal Pigmented Epithelial (hESC-RPE) Cells in Patients With Stargardt's Macular Dystrophy (SMD)
Brief Title: A Follow up Study to Determine the Safety and Tolerability of Sub-retinal Transplantation of Human Embryonic Stem Cell Derived Retinal Pigmented Epithelial (hESC-RPE) Cells in Patients With Stargardt's Macular Dystrophy (SMD)
Status: Completed | Type: Observational
Sponsor: Astellas Institute for Regenerative Medicine (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 7316-CL-0006; 2012-002827-14 (EudraCT Number); ACT-hESC-RPE-SMD-01FU EU (Other: Sponsor)
Record Dates: First submitted 2016-10-20; First posted 2016-10-21 (Estimated); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Stargardt's Macular Dystrophy
Keywords: Stargardt's Macular Dystrophy; Retinal Diseases; Macular Degeneration; fundus flavimaculatus; hESC-RPE; ASP7316; juvenile macular dystrophy; SMD
MeSH Terms: conditions — Retinal Diseases; Macular Degeneration; Stargardt Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- uniocular subretinal injection of hESC-RPE cells: Cohort 1. 50,000 cells transplanted; Cohort 2. 100,000 cells transplanted; Cohort 3. 150,000 cells transplanted; Cohort 4. 200,000 cells transplanted
  Interventions: Biological: hESC-RPE

INTERVENTIONS:
Biological: hESC-RPE — sub-retinal injection
  Other Names: ASP7316

SUMMARY:
The purpose of this study is to evaluate the long term safety and tolerability of hESC-RPE cellular therapy in patients with advanced SMD from 1 to 5 years following the surgical procedure to implant the hESC-RPE cells.

DETAILED DESCRIPTION:
This study is a long-term, follow- up of a Phase I/II, open-label, non-randomized, 4-cohort, dose escalation, multi-center clinical trial (referred to as the core trial or core protocol) in which a maximum of 12 SMD patients were transplanted with sequential doses of hESC-RPE cells, starting at a dose of 50,000 hESC-RPE cells transplanted and increasing to a maximum dose of 200,000 hESC-RPE cells transplanted. All patients who participate in the core protocol are eligible for participation in the follow-up protocol. The first visit of this extension protocol will correspond to the last visit of the core protocol, and will take place at 12 months post-cell implantation. Informed consent for this follow-up protocol will be obtained at the first visit which will occur at the 12-month visit of the core protocol. Patients will be evaluated at 18, 24, 36, 48 and 60 months post-transplant (or more frequently as clinically indicated). Follow-up will include obtaining information about ophthalmological findings and events of special interest as defined in the Primary Outcome. At the last visit of this follow up study, whether at 60 months post-transplant or at early discontinuation, patients will be invited to participate in a life-long annual health survey, under a separate protocol, to further monitor long-term safety.

ELIGIBILITY:
Inclusion Criteria:

* Must have been treated with hESC-RPE cell transplant in the core protocol.
* Able to understand and willing to sign the informed consent to participate in the follow-up study.

Exclusion Criteria:

* There are no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is by invitation only from previous participants in the core protocol.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2013-01-16 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-10-02 (Actual)

PRIMARY OUTCOMES:
Safety assessed by Adverse Events (AEs) of special interest in regards to the investigational product | 4 years
  This will include obtaining information about Serious Adverse Events (SAEs) that are neurologic, infectious, hematologic or fatal, any Adverse Event (AE) that causes the subject to withdraw from the study, any new diagnosis of an ocular or immune-mediated disorder, cancer (irrespective of prior history), ectopic or proliferative cell growth (Retinal pigment epithelium (RPE) or non-RPE) with adverse clinical consequence, unexpected, clinically significant AE possibly related to the cell transplant procedure or the investigational product (hESC-RPE cells), Pregnancy in a female subject or the partner of a male subject and pregnancy outcome.

SECONDARY OUTCOMES:
Incidence of graft failure or rejection | 4 years
  Evidence of graft failure or rejection may consist of: Presence of retinal edema, cystoid macular edema, retinal white dots, retinal hemorrhage, serous retinal detachment, sub-retinal exudates, sub-retinal fibrosis, ocular vascular and/or optic disc leakage, and elevated intraocular pressure or hypotony. Evidence of unanticipated and persistent or increasing non-infectious ocular inflammation (e.g., vasculitis, retinitis, choroiditis, vitritis, pars planitis, anterior segment inflammation/uveitis).
Number of patients with changes in ocular examinations or images | 4 years
  The number of patients with clinically significant absolute values or changes from baseline in Intra-ocular pressure (IOP) and Best Corrected Visual Acuity (BCVA) will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Institute for Regenerative Medicine
Locations (2):
- United Kingdom (2):
  - Moorefields Eye Hospital NHS Foundation Trust, London
  - Newcastle on Tyne NHS Foundation Trust, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/study.aspx?ID=394